CLINICAL TRIAL: NCT03920787
Title: Effects of Inositol Supplementation in Children With Excessive Body Weight and Insulin Resistance
Brief Title: Evaluating the Effect of Inositol Supplementation in Overweight Children on Basal Insulin and Body Weight
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Alice Andreassi (Other)
Collaborators: Lo.Li.Pharma s.r.l (Industry); Azienda Ospedaliera San Paolo (Other)
Responsible Party: Sponsor-Investigator, Alice Andreassi, Principal Investigator, Azienda Ospedaliera San Paolo
Organization: Azienda Ospedaliera San Paolo (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2017/ST/222
Record Dates: First submitted 2019-04-16; First posted 2019-04-19 (Actual); Last update posted 2019-04-22 (Actual); Status verified 2019-04

CONDITIONS: Insulin Resistance
Keywords: inositol; insulin resistance; overweight; children
MeSH Terms: conditions — Insulin Resistance; Overweight

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inositol (Experimental): Administration of Inofolic Combi (Myo-inositol 1100 mg + D-Chiro-inositol 27,6 mg + Folic Acid 400 μg - Lo.Li Pharma S.r.l.) 2 capsules every day for 1 month
  Interventions: Dietary Supplement: Inofolic Combi
- Placebo (Placebo Comparator): Administration of placebo. 2 capsules every day for 1 month
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Inofolic Combi — Myo-inositol 1100 mg + D-Chiro-inositol 27,6 mg + Folic Acid 400 μg. 2 capsules every day for 1 month.
  Arms: Inositol
Other: Placebo — 2 capsules every day for 1 month
  Arms: Placebo

SUMMARY:
Inositol in involved in the insulin pathway. In literature it has been demonstrated to improve insulin sensitivity and ovarian function in women affected by PCOS.

In a preliminary study conducted on obese children between 7 and 15 years, the investigators have demonstrated that Inositol administration (Myo-inositol 1100 mg + D-Chiro-inositol 27,6 mg + Folic Acid 400 μg) before a Glucose Oral Tolerance Test reduces the increase of insulin levels, particularly in subjects with basal insulin ≥ 15 uU/ml.

So the aim of this study is to evaluate the potential therapeutic effect of inositol, as non-pharmacologic agent, in preventing tipe II diabetes in children.

ELIGIBILITY:
Inclusion Criteria:

* 8-18 years old
* overweight or obesity
* basal insulin ≥ 20 uU/ml

Exclusion Criteria:

* pubertal delay
* hypogonadism
* hypothyroidism or hyperthyroidism
* obesity-related genetic diseases

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 23 (Estimated)
Dates: Start 2018-03-10 (Actual); Primary Completion 2020-03 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Basal Insulin | 1 month
  Evaluation of the efficacy of inositol in reducing basal insulin

SECONDARY OUTCOMES:
Body weight | 1 month
  Evaluation of the efficacy of inositol in reducing body weight

CONTACTS AND LOCATIONS:
Overall Officials: Mario Mancini, Study Director — AO San Paolo
Locations (1):
- AO San Paolo, Milan, Mi, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mancini M, Andreassi A, Salvioni M, Pelliccione F, Mantellassi G, Banderali G. Myoinositol and D-Chiro Inositol in Improving Insulin Resistance in Obese Male Children: Preliminary Data. Int J Endocrinol. 2016;2016:8720342. doi: 10.1155/2016/8720342. Epub 2016 Nov 1. PMID 27882052